CLINICAL TRIAL: NCT05574725
Title: Assessment of the Predictive Value of Outpatient Smartphone Videos in Diagnosis of Epileptic Seizures
Brief Title: Diagnostic Value of Smartphone Video in Epileptic Seizures
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed abd el Moez Eissa, Hend Mohamed Abd El Moez, Assiut University
Other Study IDs: Smartphone in epilepsy
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-08

CONDITIONS: Value of Smartphone in Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Smartphone — review of the smartphone video on patients phone by general neurologist and epileptogist each separately with comment on onquality of video using videoquality scale(10), semiology, seizure diagnosis

SUMMARY:
1. Accuracy of seizure diagnosis based on smartphone seizure semiology anaysis
2. Assess the factors that affect the diagnostic reliability of smartphone videos

DETAILED DESCRIPTION:
E pilepsy has a substantial global burden of disease.1 Diagnosis is made clinically based on a historical recount of witnessed events and a laboratory assessment. Differential diagnosis for seizures is broad. Even seasoned clinicians can be misled when individuals lack medical knowledge or pertinent terminology to accurately represent witnessed seizure behavior.2Video electroencephalogram (EEG) monitoring (VEM) is recommended when there is diagnostic uncertainty in classifying seizure type or epilepsy syndrome.3 Video EEG monitoring provides objective evidence for definitive diagnosis4 ;Additionally, VEM may not be practical for some patients because of relative infrequency of events Geographic limitations, transportation constraints, and insurance coverage may also restrict access.2,4 While VEM is the criterion standard for seizure diagnosis, web-based smartphone use has become a popular means to augment clinical practice involving seizure reporting by people with epilepsy. However, smartphone videos are not recorded in a controlled environment in which the clinicians themselves are able to define when and how each spell is to be recorded,. As such, there are issues of focus, lighting, duration, and initiation that must be considered when interpreting homemade smartphone video recordings obtained by a lay population of caregivers to evaluate people with seizures on the other hand, it has been proven that discriminating seizure's semiology is a learned skill and requires specific neurologic training 11We hypothesize that outpatient smartphone videos predictive value in patients referred for evaluation of epilepsy is variable and depends on multiple factors such as seizure semiology, and interpreting physician . on the other hand, there is no consensus on quality standards and safety recommendation of smartphone videos.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were included in the study at any age
2. provided voluntary consent, completed an HP,
3. submitted an outpatient smartphone video of their primary ictal event, underwent inpatient VEM,

Exclusion Criteria:

1. Patients were exclude, pregnant women
2. had an incomplete/absent HP, had no smartphone video,
3. did not undergo VEM, had a confirmed history of mixed epileptic and nonepileptic events (based on prior VEM), declined study participation, or did not provide informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: prospective study evaluated adult outpatient smartphone videos Study participants were outpatients referred with events that could have or could not have been epileptic seizures for elective evaluation. We prospectively collected consecutive patients who presented for evaluation of seizure-like episodes Patients who were included were those who had an interpretable smartphone video of the event in question and who eventually completed EEG-video monitoring . All patients included in the final analysis signed a consent form upon admission to the video-EEG that included an agreement statement. smartphone Videos were reviewed by general neurologist and epileptogist each separately The smartphone diagnosis was then compared to the eventual diagnosis based on the gold standard video-EEG monitoring. Each interpretation will be done blinded
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2022-10-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of the predictive value of outpatient smartphone videos in diagnosis of epileptic seizures | 1 year
  Measures of performance (accuracy, sensitivity, specificity, positive predictive value, and negative predictive value) for smartphone video-based diagnosis by general neurologist and epileptogist (the index test) were compared with those for history and physical examination and video electroencephalogram monitoring (the reference standard).

SECONDARY OUTCOMES:
Assessment of the predictive value of outpatient smartphone videos in diagnosis of epileptic seizures | 1year
  descriptive analysis of factors affecting quality of smartphone videos

CONTACTS AND LOCATIONS:
Overall Officials: Hend Mohamed Abd El moez, Principal Investigator — Assiut University

REFERENCES:
- [Background] GBD 2013 DALYs and HALE Collaborators; Murray CJ, Barber RM, Foreman KJ, Abbasoglu Ozgoren A, Abd-Allah F, Abera SF, Aboyans V, Abraham JP, Abubakar I, Abu-Raddad LJ, Abu-Rmeileh NM, Achoki T, Ackerman IN, Ademi Z, Adou AK, Adsuar JC, Afshin A, Agardh EE, Alam SS, Alasfoor D, Albittar MI, Alegretti MA, Alemu ZA, Alfonso-Cristancho R, Alhabib S, Ali R, Alla F, Allebeck P, Almazroa MA, Alsharif U, Alvarez E, Alvis-Guzman N, Amare AT, Ameh EA, Amini H, Ammar W, Anderson HR, Anderson BO, Antonio CA, Anwari P, Arnlov J, Arsic Arsenijevic VS, Artaman A, Asghar RJ, Assadi R, Atkins LS, Avila MA, Awuah B, Bachman VF, Badawi A, Bahit MC, Balakrishnan K, Banerjee A, Barker-Collo SL, Barquera S, Barregard L, Barrero LH, Basu A, Basu S, Basulaiman MO, Beardsley J, Bedi N, Beghi E, Bekele T, Bell ML, Benjet C, Bennett DA, Bensenor IM, Benzian H, Bernabe E, Bertozzi-Villa A, Beyene TJ, Bhala N, Bhalla A, Bhutta ZA, Bienhoff K, Bikbov B, Biryukov S, Blore JD, Blosser CD, Blyth FM, Bohensky MA, Bolliger IW, Bora Basara B, Bornstein NM, Bose D, Boufous S, Bourne RR, Boyers LN, Brainin M, Brayne CE, Brazinova A, Breitborde NJ, Brenner H, Briggs AD, Brooks PM, Brown JC, Brugha TS, Buchbinder R, Buckle GC, Budke CM, Bulchis A, Bulloch AG, Campos-Nonato IR, Carabin H, Carapetis JR, Cardenas R, Carpenter DO, Caso V, Castaneda-Orjuela CA, Castro RE, Catala-Lopez F, Cavalleri F, Cavlin A, Chadha VK, Chang JC, Charlson FJ, Chen H, Chen W, Chiang PP, Chimed-Ochir O, Chowdhury R, Christensen H, Christophi CA, Cirillo M, Coates MM, Coffeng LE, Coggeshall MS, Colistro V, Colquhoun SM, Cooke GS, Cooper C, Cooper LT, Coppola LM, Cortinovis M, Criqui MH, Crump JA, Cuevas-Nasu L, Danawi H, Dandona L, Dandona R, Dansereau E, Dargan PI, Davey G, Davis A, Davitoiu DV, Dayama A, De Leo D, Degenhardt L, Del Pozo-Cruz B, Dellavalle RP, Deribe K, Derrett S, Des Jarlais DC, Dessalegn M, Dharmaratne SD, Dherani MK, Diaz-Torne C, Dicker D, Ding EL, Dokova K, Dorsey ER, Driscoll TR, Duan L, Duber HC, Ebel BE, Edmond KM, Elshrek YM, Endres M, Ermakov SP, Erskine HE, Eshrati B, Esteghamati A, Estep K, Faraon EJ, Farzadfar F, Fay DF, Feigin VL, Felson DT, Fereshtehnejad SM, Fernandes JG, Ferrari AJ, Fitzmaurice C, Flaxman AD, Fleming TD, Foigt N, Forouzanfar MH, Fowkes FG, Paleo UF, Franklin RC, Furst T, Gabbe B, Gaffikin L, Gankpe FG, Geleijnse JM, Gessner BD, Gething P, Gibney KB, Giroud M, Giussani G, Gomez Dantes H, Gona P, Gonzalez-Medina D, Gosselin RA, Gotay CC, Goto A, Gouda HN, Graetz N, Gugnani HC, Gupta R, Gupta R, Gutierrez RA, Haagsma J, Hafezi-Nejad N, Hagan H, Halasa YA, Hamadeh RR, Hamavid H, Hammami M, Hancock J, Hankey GJ, Hansen GM, Hao Y, Harb HL, Haro JM, Havmoeller R, Hay SI, Hay RJ, Heredia-Pi IB, Heuton KR, Heydarpour P, Higashi H, Hijar M, Hoek HW, Hoffman HJ, Hosgood HD, Hossain M, Hotez PJ, Hoy DG, Hsairi M, Hu G, Huang C, Huang JJ, Husseini A, Huynh C, Iannarone ML, Iburg KM, Innos K, Inoue M, Islami F, Jacobsen KH, Jarvis DL, Jassal SK, Jee SH, Jeemon P, Jensen PN, Jha V, Jiang G, Jiang Y, Jonas JB, Juel K, Kan H, Karch A, Karema CK, Karimkhani C, Karthikeyan G, Kassebaum NJ, Kaul A, Kawakami N, Kazanjan K, Kemp AH, Kengne AP, Keren A, Khader YS, Khalifa SE, Khan EA, Khan G, Khang YH, Kieling C, Kim D, Kim S, Kim Y, Kinfu Y, Kinge JM, Kivipelto M, Knibbs LD, Knudsen AK, Kokubo Y, Kosen S, Krishnaswami S, Kuate Defo B, Kucuk Bicer B, Kuipers EJ, Kulkarni C, Kulkarni VS, Kumar GA, Kyu HH, Lai T, Lalloo R, Lallukka T, Lam H, Lan Q, Lansingh VC, Larsson A, Lawrynowicz AE, Leasher JL, Leigh J, Leung R, Levitz CE, Li B, Li Y, Li Y, Lim SS, Lind M, Lipshultz SE, Liu S, Liu Y, Lloyd BK, Lofgren KT, Logroscino G, Looker KJ, Lortet-Tieulent J, Lotufo PA, Lozano R, Lucas RM, Lunevicius R, Lyons RA, Ma S, Macintyre MF, Mackay MT, Majdan M, Malekzadeh R, Marcenes W, Margolis DJ, Margono C, Marzan MB, Masci JR, Mashal MT, Matzopoulos R, Mayosi BM, Mazorodze TT, Mcgill NW, Mcgrath JJ, Mckee M, Mclain A, Meaney PA, Medina C, Mehndiratta MM, Mekonnen W, Melaku YA, Meltzer M, Memish ZA, Mensah GA, Meretoja A, Mhimbira FA, Micha R, Miller TR, Mills EJ, Mitchell PB, Mock CN, Mohamed Ibrahim N, Mohammad KA, Mokdad AH, Mola GL, Monasta L, Montanez Hernandez JC, Montico M, Montine TJ, Mooney MD, Moore AR, Moradi-Lakeh M, Moran AE, Mori R, Moschandreas J, Moturi WN, Moyer ML, Mozaffarian D, Msemburi WT, Mueller UO, Mukaigawara M, Mullany EC, Murdoch ME, Murray J, Murthy KS, Naghavi M, Naheed A, Naidoo KS, Naldi L, Nand D, Nangia V, Narayan KM, Nejjari C, Neupane SP, Newton CR, Ng M, Ngalesoni FN, Nguyen G, Nisar MI, Nolte S, Norheim OF, Norman RE, Norrving B, Nyakarahuka L, Oh IH, Ohkubo T, Ohno SL, Olusanya BO, Opio JN, Ortblad K, Ortiz A, Pain AW, Pandian JD, Panelo CI, Papachristou C, Park EK, Park JH, Patten SB, Patton GC, Paul VK, Pavlin BI, Pearce N, Pereira DM, Perez-Padilla R, Perez-Ruiz F, Perico N, Pervaiz A, Pesudovs K, Peterson CB, Petzold M, Phillips MR, Phillips BK, Phillips DE, Piel FB, Plass D, Poenaru D, Polinder S, Pope D, Popova S, Poulton RG, Pourmalek F, Prabhakaran D, Prasad NM, Pullan RL, Qato DM, Quistberg DA, Rafay A, Rahimi K, Rahman SU, Raju M, Rana SM, Razavi H, Reddy KS, Refaat A, Remuzzi G, Resnikoff S, Ribeiro AL, Richardson L, Richardus JH, Roberts DA, Rojas-Rueda D, Ronfani L, Roth GA, Rothenbacher D, Rothstein DH, Rowley JT, Roy N, Ruhago GM, Saeedi MY, Saha S, Sahraian MA, Sampson UK, Sanabria JR, Sandar L, Santos IS, Satpathy M, Sawhney M, Scarborough P, Schneider IJ, Schottker B, Schumacher AE, Schwebel DC, Scott JG, Seedat S, Sepanlou SG, Serina PT, Servan-Mori EE, Shackelford KA, Shaheen A, Shahraz S, Shamah Levy T, Shangguan S, She J, Sheikhbahaei S, Shi P, Shibuya K, Shinohara Y, Shiri R, Shishani K, Shiue I, Shrime MG, Sigfusdottir ID, Silberberg DH, Simard EP, Sindi S, Singh A, Singh JA, Singh L, Skirbekk V, Slepak EL, Sliwa K, Soneji S, Soreide K, Soshnikov S, Sposato LA, Sreeramareddy CT, Stanaway JD, Stathopoulou V, Stein DJ, Stein MB, Steiner C, Steiner TJ, Stevens A, Stewart A, Stovner LJ, Stroumpoulis K, Sunguya BF, Swaminathan S, Swaroop M, Sykes BL, Tabb KM, Takahashi K, Tandon N, Tanne D, Tanner M, Tavakkoli M, Taylor HR, Te Ao BJ, Tediosi F, Temesgen AM, Templin T, Ten Have M, Tenkorang EY, Terkawi AS, Thomson B, Thorne-Lyman AL, Thrift AG, Thurston GD, Tillmann T, Tonelli M, Topouzis F, Toyoshima H, Traebert J, Tran BX, Trillini M, Truelsen T, Tsilimbaris M, Tuzcu EM, Uchendu US, Ukwaja KN, Undurraga EA, Uzun SB, Van Brakel WH, Van De Vijver S, van Gool CH, Van Os J, Vasankari TJ, Venketasubramanian N, Violante FS, Vlassov VV, Vollset SE, Wagner GR, Wagner J, Waller SG, Wan X, Wang H, Wang J, Wang L, Warouw TS, Weichenthal S, Weiderpass E, Weintraub RG, Wenzhi W, Werdecker A, Westerman R, Whiteford HA, Wilkinson JD, Williams TN, Wolfe CD, Wolock TM, Woolf AD, Wulf S, Wurtz B, Xu G, Yan LL, Yano Y, Ye P, Yentur GK, Yip P, Yonemoto N, Yoon SJ, Younis MZ, Yu C, Zaki ME, Zhao Y, Zheng Y, Zonies D, Zou X, Salomon JA, Lopez AD, Vos T. Global, regional, and national disability-adjusted life years (DALYs) for 306 diseases and injuries and healthy life expectancy (HALE) for 188 countries, 1990-2013: quantifying the epidemiological transition. Lancet. 2015 Nov 28;386(10009):2145-91. doi: 10.1016/S0140-6736(15)61340-X. Epub 2015 Aug 28. PMID 26321261
- [Background] Deacon C, Wiebe S, Blume WT, McLachlan RS, Young GB, Matijevic S. Seizure identification by clinical description in temporal lobe epilepsy: how accurate are we? Neurology. 2003 Dec 23;61(12):1686-9. doi: 10.1212/01.wnl.0000090566.40544.04. PMID 14694030
- [Background] Velis D, Plouin P, Gotman J, da Silva FL; ILAE DMC Subcommittee on Neurophysiology. Recommendations regarding the requirements and applications for long-term recordings in epilepsy. Epilepsia. 2007 Feb;48(2):379-84. doi: 10.1111/j.1528-1167.2007.00920.x. PMID 17295634
- [Background] Cascino GD. Clinical indications and diagnostic yield of video-electroencephalographic monitoring in patients with seizures and spells. Mayo Clin Proc. 2002 Oct;77(10):1111-20. doi: 10.4065/77.10.1111. PMID 12374255
- [Background] Goldenholz DM, Moss R, Jost DA, Crone NE, Krauss G, Picard R, Caborni C, Cavazos JE, Hixson J, Loddenkemper T, Salazar TD, Lubbers L, Harte-Hargrove LC, Whittemore V, Duun-Henriksen J, Dolan E, Kasturia N, Oberemk M, Cook MJ, Lehmkuhle M, Sperling MR, Shafer PO. Common data elements for epilepsy mobile health systems. Epilepsia. 2018 May;59(5):1020-1026. doi: 10.1111/epi.14066. Epub 2018 Mar 31. PMID 29604050